CLINICAL TRIAL: NCT05653921
Title: Prospective Study to Validate the Imaging Biomarker for Neuropathic Corneal Pain.
Brief Title: Prospective Study to Validate the Imaging Biomarker for NCP (R33)
Status: Suspended | Type: Observational
Why Stopped: PI si leaving institution. This study will likely be transferred to USF but study activity is not continuing at TMC.
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: STUDY00003018; 4R33NS113341-02 (NIH)
Record Dates: First submitted 2022-09-06; First posted 2022-12-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Syndromes; Corneal Disease
MeSH Terms: conditions — Dry Eye Syndromes; Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dry Eye Disease Group: Symptoms of ocular surface discomfort or dry eye disease for at least 3 months, supported by clinical exam findings. Reported quality of life is not effected by ocular pain.
  Interventions: Other: In vivo confocal microscopy (IVCM)
- Neuropathic Corneal Pain Group: Symptoms of ocular surface discomfort or pain for at least 3 months, that are reported to have a significant impact on quality of life and ability to perform daily activities.
  Interventions: Other: In vivo confocal microscopy (IVCM)
- Control Group: No symptoms of ocular surface discomfort or dry eye disease.
  Interventions: Other: In vivo confocal microscopy (IVCM)

INTERVENTIONS:
Other: In vivo confocal microscopy (IVCM) — In vivo confocal microscopy (IVCM) allows for visualization of the corneal structures at the cellular level, allowing for assessment of corneal nerves. With a magnification of 800 times, it makes it possible to detect and quantify changes in the epithelial layers and sub-basal nerve plexus.

SUMMARY:
The aim of this study is establish the reliability and clinical utility of microneuromas as identified via in vivo confocal microscopy as the diagnostic biomarker for NCP.

DETAILED DESCRIPTION:
Dry Eye Disease (DED) is a multifactorial disease of the ocular surface characterized by a loss of homeostasis of the tear film, and accompanied by ocular symptoms, in which tear film instability and hyperosmolarity, ocular surface inflammation and damage, and neurosensory abnormalities.

Neuropathic corneal pain (NCP), an ocular and severe type of neuropathic pain describes patients with symptoms of ocular discomfort out of proportion with clinical signs. The lack of clinical signs observed by standard ophthalmic examination has resulted in underdiagnosis of NCP or misdiagnosis as dry eye disease. Thus, having a biomarker for NCP is critical to identify and treat these patients. No biomarker or clinical signs exists to identify NCP patients.

Investigating corneal neurosensory abnormalities could help to diagnose NCP and potentially differentiate these patients from those with DED. In vivo confocal microscopy (IVCM) allows for real-time optical biopsies at a quasi-histological level, allowing for assessment of corneal nerves. IVCM non-invasive diagnostic imaging across NCP, DED, and healthy individuals will be analyzed to validate corneal microneuromas as a biomarker for NCP.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

1. 18 years of age or older
2. Ability to consent
3. Best corrected visual acuity of 20/40 or better in each eye

Dry Eye Disease Group:

1. Chief complaint is ocular surface discomfort or dry eye disease, but subject reports no ocular pain on OPAS questionnaire
2. Symptoms lasting at least 3 months
3. Presence of at least two of the following within the same eye:

   1. Anesthetized Schirmer score =/< 10mm
   2. Corneal staining of >3/15 based on NEI scale
   3. Tear break up time < 10 seconds

Neuropathic Corneal Pain Group:

1. Chief complain is ocular surface discomfort or dry eye disease
2. Symptoms lasting at least 3 months
3. All of the following in both eyes:

   1. Corneal staining of less than or equal to 3/15 based on NEI scale
   2. Tear break up time =/> 10 seconds
4. Must have at least 25% peripheral pain
5. Subject reported discomfort prior to drop response testing of at least 3 out of 10

Control Group:

1. No symptoms of ocular surface discomfort or dry eye disease
2. All of the following in both eyes

   1. Anesthetized Schirmer score > 10 mm
   2. Corneal staining of less than or equal to 3/15 based on NEI scale
   3. Tear break up time > 10 seconds
3. The same sex and within 5 years of age of a patient within the NCP group.

Exclusion Criteria:

1. Pregnant or nursing
2. Irregular corneal disease
3. Ocular surgery in the past 3 months
4. Ocular infection in the past 3 months
5. Active ocular allergies
6. Participation in a study that could potentially impact the IVCM in the opinion of the investigator
7. Current use of corneal nerve regeneration therapy that has been on-going for 3 months or more.
8. For NCP group only, patients for whom their pain and symptoms can be attributed to other causes in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will not be limiting the inclusion of the NCP or DED groups for this study. We will be recruiting from two Cornea Clinics in diverse large cities of Boston and Philadelphia. Thus, the sample collected from this group is expected to be representative of the population for each of these groups. We will be limiting inclusion of the control group to those age and sex matched controls as described above. This will allow for the conclusions drawn from this study to be more applicable in clinical practice. Without an age and sex matched control group, one could attribute differences in IVCM to these two variables instead of the disease(s).
Sampling Method: Non-Probability Sample
Enrollment: 438 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Presence of microneuromas as assessed by in vivo confocal microscopy (IVCM). | Day 1
  The obtained sequence of IVCM imaging scans of both eyes will be evaluated for findings of microneuromas; defined as either observed presence or absence of microneuroma

SECONDARY OUTCOMES:
Intra-subject repeatability; Presence of the microneuroma biomarker in the same participant at 2 weeks | From Day 1 to 2 weeks
  Confirmation of presence of microneuroma on IVCM at 2 weeks in participants with IVCM finding of microneruoma at Visit 1
Establish the reference interval for the microneuroma biomarker | Day 1
  Quantification of microneuromas as assessed by IVCM in each cohort (Normal vs. NCP vs. DED)
Ocular Pain Assessment Survey (OPAS) questionnaire results correlation to microneuromas; OPAS reported quality of life score compared across the 3 cohorts. | Day 1
  Ocular Pain Assessment Survey (OPAS) questionnaire: 27-item quantitative questionnaire designed to provide an assessment of the symptoms and quality of life effect of ocular pain. The 27 items of the OPAS questionnaire are graded on a scale of 0 to 10, or 10 to 100, where 0 indicates none and 10 or 100 indicate maximum. Higher scores indicate greater impact of ocular pain on quality of life dimensions.
Hyperosmolar functional nerve tests in correlation to microneuromas; hyperosmolar functional nerve tests results compared cross cohorts | Day 1
  Using the Pain Visual Analogue Scale (VAS), Symptoms of ocular comfort and dryness at the time in question will be graded for each eye verbally on a scale of 0-10, where 0=excellent comfort, no dryness and 10=extremely uncomfortable, extremely dry. A single drop of hypertonic sodium chloride solution (Muro 128®, 5%) at room temperature will be instilled into each eye. After 20 seconds, participants will be asked to grade their ocular comfort and dryness symptoms as described in the VAS procedure again allowing assessment of changes in sensation due to the hyperosmolar drop and activation of the polymodal nociceptors
Test the utility of already configured AI software to diagnose NCP patients | Day 1 to 2 weeks
  categorical variables of NCP and DED as diagnosed by the AI system and the classification of subjects into the NCP and DED groups based on inclusion criteria set by the study

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — Tufts Medical Center
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iuganov EM, Krylov IuV, Kuznetsov VS. [Use of psychophysiological indices in the practice of audiological studies]. Izv Akad Nauk SSSR Biol. 1971 Jul-Aug;4:587-95. No abstract available. Russian. PMID 5121784
- [Background] Fry HJ. Overuse syndrome, alias tenosynovitis/tendinitis: the terminological hoax. Plast Reconstr Surg. 1986 Sep;78(3):414-7. doi: 10.1097/00006534-198609000-00025. No abstract available. PMID 3737766
- [Background] Nichols KK, Nichols JJ, Mitchell GL. The lack of association between signs and symptoms in patients with dry eye disease. Cornea. 2004 Nov;23(8):762-70. doi: 10.1097/01.ico.0000133997.07144.9e. PMID 15502475
- [Background] Sullivan BD, Crews LA, Messmer EM, Foulks GN, Nichols KK, Baenninger P, Geerling G, Figueiredo F, Lemp MA. Correlations between commonly used objective signs and symptoms for the diagnosis of dry eye disease: clinical implications. Acta Ophthalmol. 2014 Mar;92(2):161-6. doi: 10.1111/aos.12012. Epub 2012 Dec 28. PMID 23279964
- [Background] Nichols KK, Bacharach J, Holland E, Kislan T, Shettle L, Lunacsek O, Lennert B, Burk C, Patel V. Impact of Dry Eye Disease on Work Productivity, and Patients' Satisfaction With Over-the-Counter Dry Eye Treatments. Invest Ophthalmol Vis Sci. 2016 Jun 1;57(7):2975-82. doi: 10.1167/iovs.16-19419. PMID 27273596
- [Background] Fovaeus M, Andersson KE, Hedlund H. Calcium channel blockade and contractile responses in the isolated human vas deferens. J Urol. 1987 Sep;138(3):654-8. doi: 10.1016/s0022-5347(17)43292-7. PMID 2442424
- [Background] Classification of Chronic Pain, Part III: Pain Terms, A Current List with Definitions and Notes on Usage. Second ed. Seattle: IASP Press; 1994
- [Background] Dieckmann G, Koseoglu N, Moein HR, Kataguiri P, Hamrah P. Epidemiological factors of neuropathic corneal pain. IASP: The 18th World Congress on Pain; 2018; Boston, MA.
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Yu J, Asche CV, Fairchild CJ. The economic burden of dry eye disease in the United States: a decision tree analysis. Cornea. 2011 Apr;30(4):379-87. doi: 10.1097/ICO.0b013e3181f7f363. PMID 21045640
- [Background] Lopez MJ, Jamali A, Dieckmann G, et al. Corneal Pain Has a Negative Impact on the Quality of Life of Patients with Neuropathic Corneal Pain. Investigative ophthalmology & visual science. 2018;59(9):138-138
- [Background] Lopez MJ, Abbouda A, Pondelis N, et al. The Ocular Pain Assessment Survey and In Vivo Confocal Microscopy as Valuable Tools in the Diagnosis and Management of Patients with Corneal Neuropathic Pain. Investigative ophthalmology & visual science. 2017;58(8):1013-1013.